CLINICAL TRIAL: NCT01005160
Title: A Sequence-randomized, Open-label, Multiple Dosing, Three-way Crossover Clinical Trial to Investigate the Pharmacokinetic Drug Interaction Between CKD-501 and Metformin After Oral Administration in Healthy Male Volunteers
Brief Title: Drug Interaction Between CKD-501 and Metformin
Acronym: CKD-19HPS09H
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Chin Kim, Chong Kun Dang
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CKD-19HPS09H; 19HPS09H
Record Dates: First submitted 2009-10-28; First posted 2009-10-30 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2009-10

CONDITIONS: Healthy Male Volunteers
Keywords: Mellitus, type 2; pharmacokinetic evaluation; drug interaction between CKD-501 and metformin
MeSH Terms: interventions — Metformin; lobeglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CKD501 (Experimental)
  Interventions: Drug: Metformin; Drug: CKD-501

INTERVENTIONS:
Drug: Metformin — CKD-501 0.5mg, metformin 1000mg
  Other Names: Lobeglitazone
Drug: CKD-501 — CKD-501 0.5mg, metformin 1000mg
  Other Names: Lobeglitazone

SUMMARY:
The purpose of this study is to evaluate safety, tolerance by comparing availability and the pharmacokinetic drug interaction between the CKD-501 and metformin when administered alone and combination to healthy male volunteers.

DETAILED DESCRIPTION:
Volunteers doses three times over the period of CKD-501 0.5mg and metformin 1000mg alone, repeated doses are five days.

In addition, the CKD-501 0.5mg and metformin 1000mg are administered simultaneously be used repeatedly to five days.

Every time before and after each medication safety and drug absorption, distribution, metabolism and excretion rate, and is expected to conduct some tests.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 aged and 45 aged in healthy males
* Weight more than 55kg, IBW 20% within the range
* FPG 70~125 mg/dL
* Agreement with written informed consent

Exclusion Criteria:

* Clinically significant disease(liver, heart, immune system, Respiratory system, Endocrine system, blood tumor disease, Mental illness)or a history that has learned
* Test drug may affect the absorption of the gastrointestinal disease or a history that has learned
* Hypersensitivity reactions to drugs or Clinically significant hypersensitivity reactions in the history of party
* AST, ALT level over to 1.5 times and creatinine clearance less 80mL/min
* systolic blood pressure less than 100mmHg or 150mmHg, diastolic blood pressure less than 60mmHg or greater than 95mmHg
* Substance abuse, or a history of drug abuse showed a positive for the party
* Medication within 2 weeks in the first professional medical, medicine, OTC, vitamins taking
* Previously participated in other trial within 2 months
* Medication within 2 months make whole blood donation or medication within 1 month in component blood donation
* Continued to be drunk or during clinical trials can not be drunk
* 10 cigarettes a day for the last 3 months than the average smoker or during clinical trials can not be smoke
* Containing grapefruit foods ingested during clinical trials or can not be ingested
* Containing caffeine foods ingested during 24 hours before admission to hospital of can not be ingested

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
CKD - 501 and metformin Pharmacokinetics evaluation | 16 days

SECONDARY OUTCOMES:
CKD-501 and metformin safety evaluation | 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Kyung S Yu, Principal Investigator — Seoul National University Hospital

REFERENCES:
- [Derived] Shin D, Kim TE, Yoon SH, Cho JY, Shin SG, Jang IJ, Yu KS. Assessment of the pharmacokinetics of co-administered metformin and lobeglitazone, a thiazolidinedione antihyperglycemic agent, in healthy subjects. Curr Med Res Opin. 2012 Jul;28(7):1213-20. doi: 10.1185/03007995.2012.703131. Epub 2012 Jul 2. PMID 22697273